CLINICAL TRIAL: NCT05441878
Title: To Compare 20% Albumin vs. Balanced Salt Solution as Resuscitation Fluid and Identify Fluid Responsiveness Criteria in Critically Ill Patients With Cirrhosis With Sepsis Induced Hypotension; a Prospective Randomized Controlled Trial.
Brief Title: 20% Albumin vs. Balanced Salt Solution as Resuscitation Fluid in Cirrhosis With Sepsis Induced Hypotension
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Madhumita Premkumar, Assistant professor, Department of Hepatology, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IEC/11/2019/1496
Record Dates: First submitted 2022-04-26; First posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Cirrhosis, Liver; Acute-On-Chronic Liver Failure; Shock, Septic; Shock Hypovolemic
MeSH Terms: conditions — Liver Cirrhosis; Acute-On-Chronic Liver Failure; Shock, Septic; Shock | interventions — Albumins; Hanks Balanced Salt Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 20% Albumin arm (Experimental): 20% Albumin in a dose of 20-40 gm per day as infusion over 12-24 h
  Interventions: Drug: 20% albumin; Drug: Balanced salt solution
- Balanced salt solution arm (Active Comparator): Fluid resuscitation protocol includes use of an immediate 500 ml bolus of crystalloid i.e., balanced salt solution (BSS) or 0.9% normal saline (Rescue phase), followed by 20 ml/kg fluid in the first 6 hours titrated to target MAP of > 65mmHg.The second phase of fluid resuscitation (Optimization phase) will be performed as per IVC targets, attainment of lactate clearance, and LUS score to prevent overload.
  Interventions: Drug: Balanced salt solution

INTERVENTIONS:
Drug: 20% albumin — Albumin arm for resuscitation fluid
  Arms: 20% Albumin arm
Drug: Balanced salt solution — Only Balanced salt solution will be used.

SUMMARY:
Patients with cirrhosis patients have a high incidence of sepsis which can trigger decompensation and may result in prolonged hospital stay and increased mortality. About 30%-50% admissions of patients with cirrhosis have sepsis at presentation and about 15% patients admitted to hospital develop sepsis during the hospital stay . After infection develops, the patient may develop acute kidney injury (AKI), shock, encephalopathy or disseminated intravascular coagulation (DIC) further decreasing the chances of survival. In fact, sepsis in patients with cirrhosis is associated with 15% in-hospital mortality, approximately double that of patients without sepsis. So, sepsis is directly responsible for 30-50% of deaths in cirrhosis . Therefore, it is critical to manage sepsis early and appropriately in cirrhosis to reduce the complications and mortality. Early administration of fluids, source control and empirical antibiotics along with vasopressors if refractory shock are essential components of treatment in all patients with sepsis. Currently, the most accepted strategy for early sepsis management is a combination of early goal directed therapy (EGDT) and physiological parameters, such as urine output, lactate clearance, and administration of antibiotics, within 1 hour of presentation . The use of central venous pressure assessment is fallacious for gauging adequacy of fluid resuscitation in cirrhosis, and the difficulty of performing echocardiographic assessments in the setting of ascites and cirrhotic cardiomyopathy is also well described .

ELIGIBILITY:
Inclusion Criteria:

* Clinical/Imaging or Biopsy proven liver cirrhosis of any etiology who consent for enrolment.
* Hypotension (Mean arterial pressure <65mmHg or Systolic blood pressure <90mmHg)
* Aged between18-65 yrs

Exclusion Criteria:

* Already received colloid or more than 2 litres of fluid without baseline echocardiographic assessment.
* Already on vasopressors/inotropes
* Severe pre-existing cardiopulmonary disease
* Acute Respiratory Distress Syndrome (ARDS)
* Active bleeding like variceal bleed
* Cerebrovascular events
* Chronic renal disease - End Stage Renal Disease (ESRD)/ patient on renal replacement therapy
* Admission to ICU following liver transplantation, burns, cardiac surgery
* Brain death or likely brain death within 24 hours
* Previous adverse reaction to human albumin solution
* Pregnant or lactating women
* Informed consent refused by patient or attendants

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-08-15 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
To compare the efficacy of 20% Albumin vs Plasmalyte in the first 3 -6 hours of volume resuscitation in cirrhosis with sepsis induced hypotension and assess IVC dynamics. | At enrolment
  To compare the IVC dynamics in patients with cirrhosis and sepsis induced hypotension
To compare the efficacy of 20% Albumin vs Plasmalyte in the first 3 -6 hours of volume resuscitation in cirrhosis with sepsis induced hypotension and assess IVC dynamics. | At 6 hours
  To compare the IVC dynamics in patients with cirrhosis and sepsis induced hypotension
To compare the efficacy of 20% Albumin vs Plasmalyte in the first 3 -6 hours of volume resuscitation in cirrhosis with sepsis induced hypotension and assess IVC dynamics. | At 24 hours
  To compare the IVC dynamics in patients with cirrhosis and sepsis induced hypotension
To compare the efficacy of 20% Albumin vs Plasmalyte in the first 3 -6 hours of volume resuscitation in cirrhosis with sepsis induced hypotension and assess IVC dynamics. | At 48 hours.
  To compare the IVC dynamics in patients with cirrhosis and sepsis induced hypotension
To compare the efficacy of 20% Albumin vs Plasmalyte in the first 3 -6 hours of volume resuscitation in cirrhosis with sepsis induced hypotension and assess dynamic changes in cardiac output, stroke volume and E/e' echocardiographic parameters. | At enrolment
  To compare the cardiac output in patients with cirrhosis and sepsis induced hypotension
To compare the efficacy of 20% Albumin vs Plasmalyte in the first 3 -6 hours of volume resuscitation in cirrhosis with sepsis induced hypotension and assess dynamic changes in cardiac output, stroke volume and E/e' echocardiographic parameters. | At 24 hours
  To compare the cardiac output in patients with cirrhosis and sepsis induced hypotension
To compare the efficacy of 20% Albumin vs Plasmalyte in the first 3 -6 hours of volume resuscitation in cirrhosis with sepsis induced hypotension and assess dynamic changes in cardiac output, stroke volume and E/e' echocardiographic parameters. | At 48 hours.
  To compare the cardiac output in patients with cirrhosis and sepsis induced hypotension
To compare the efficacy of 20% Albumin vs Plasmalyte in the first 3 -6 hours of volume resuscitation in cirrhosis with sepsis induced hypotension and assess new onset of hepatorenal syndrome (HRS) or acute kidney injury (AKI) | At enrolment
  To compare the new onset of hepatorenal syndrome (HRS) or acute kidney injury (AKI)in patients with cirrhosis and sepsis induced hypotension
To compare the efficacy of 20% Albumin vs Plasmalyte in the first 3 -6 hours of volume resuscitation in cirrhosis with sepsis induced hypotension and assess new onset of hepatorenal syndrome (HRS) or acute kidney injury (AKI) | At 48 hours.
  To compare the new onset of hepatorenal syndrome (HRS) or acute kidney injury (AKI)in patients with cirrhosis and sepsis induced hypotension

SECONDARY OUTCOMES:
Urinary marker of AKI (NGal) | At enrolment
Change in urinary markers of AKI (NGal) | At 24 hours.
Change in urinary markers of AKI(NGal) | At 48 hours.
To compare the efficacy of 20% Albumin vs Plasmalyte in the first 3 -6 hours of volume resuscitation in cirrhosis with sepsis induced hypotension., and assess vasopressor requirement | At enrolment
  To compare the vasopressor requirement in patients with cirrhosis and sepsis induced hypotension
To compare the efficacy of 20% Albumin vs Plasmalyte in the first 3 -6 hours of volume resuscitation in cirrhosis with sepsis induced hypotension., and assess vasopressor requirement | At 24 hours
  To compare the vasopressor requirement in patients with cirrhosis and sepsis induced hypotension

CONTACTS AND LOCATIONS:
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, India

REFERENCES:
- [Background] Borzio M, Salerno F, Piantoni L, Cazzaniga M, Angeli P, Bissoli F, Boccia S, Colloredo-Mels G, Corigliano P, Fornaciari G, Marenco G, Pistara R, Salvagnini M, Sangiovanni A. Bacterial infection in patients with advanced cirrhosis: a multicentre prospective study. Dig Liver Dis. 2001 Jan-Feb;33(1):41-8. doi: 10.1016/s1590-8658(01)80134-1. PMID 11303974
- [Background] Navasa M, Fernandez J, Rodes J. Bacterial infections in liver cirrhosis. Ital J Gastroenterol Hepatol. 1999 Oct;31(7):616-25. PMID 10604106
- [Background] Wong F, Bernardi M, Balk R, Christman B, Moreau R, Garcia-Tsao G, Patch D, Soriano G, Hoefs J, Navasa M; International Ascites Club. Sepsis in cirrhosis: report on the 7th meeting of the International Ascites Club. Gut. 2005 May;54(5):718-25. doi: 10.1136/gut.2004.038679. PMID 15831923
- [Background] Moreau R, Hadengue A, Soupison T, Kirstetter P, Mamzer MF, Vanjak D, Vauquelin P, Assous M, Sicot C. Septic shock in patients with cirrhosis: hemodynamic and metabolic characteristics and intensive care unit outcome. Crit Care Med. 1992 Jun;20(6):746-50. doi: 10.1097/00003246-199206000-00008. PMID 1597026
- [Background] ARISE Investigators; ANZICS Clinical Trials Group; Peake SL, Delaney A, Bailey M, Bellomo R, Cameron PA, Cooper DJ, Higgins AM, Holdgate A, Howe BD, Webb SA, Williams P. Goal-directed resuscitation for patients with early septic shock. N Engl J Med. 2014 Oct 16;371(16):1496-506. doi: 10.1056/NEJMoa1404380. Epub 2014 Oct 1. PMID 25272316
- [Background] Mouncey PR, Osborn TM, Power GS, Harrison DA, Sadique MZ, Grieve RD, Jahan R, Harvey SE, Bell D, Bion JF, Coats TJ, Singer M, Young JD, Rowan KM; ProMISe Trial Investigators. Trial of early, goal-directed resuscitation for septic shock. N Engl J Med. 2015 Apr 2;372(14):1301-11. doi: 10.1056/NEJMoa1500896. Epub 2015 Mar 17. PMID 25776532
- [Background] Marik PE, Baram M, Vahid B. Does central venous pressure predict fluid responsiveness? A systematic review of the literature and the tale of seven mares. Chest. 2008 Jul;134(1):172-8. doi: 10.1378/chest.07-2331. PMID 18628220